CLINICAL TRIAL: NCT00006086
Title: Phase I Study of BMS-188797 in Combination With Carboplatin in Patients With Advanced Malignancies
Brief Title: BMS-188797 and Carboplatin in Treating Patients With Advanced Nonhematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068078; MCC-12176; BMS-CA159-003; NCI-G00-1825
Record Dates: First submitted 2000-08-03; First posted 2003-05-22 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2002-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — BMS188797; Carboplatin

INTERVENTIONS:
Drug: BMS-188797
Drug: carboplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of BMS-188797 and carboplatin in treating patients who have advanced nonhematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the recommended phase II dose based on the maximum tolerated dose of BMS-188797 when administered with carboplatin in patients with advanced nonhematologic malignancies.
* Assess the dose limiting toxicities and safety of this treatment regimen in these patients.
* Determine the plasma pharmacokinetics of this treatment regimen in these patients.
* Determine any antitumor activity of this treatment regimen in these patients.

OUTLINE: This is a dose escalation study of BMS-188797.

Patients receive BMS-188797 IV over 1 hour followed by carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of BMS-188797 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 6 patients experience dose limiting toxicities.

Patients are followed for 4 weeks, and then every 3 months thereafter.

PROJECTED ACCRUAL: Approximately 35 patients will be accrued for this study over 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced nonhematologic malignancy that has progressed on standard therapy or for which no curative therapy exists
* No brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* ALT and AST no greater than 2.5 times upper limit of normal (ULN) unless due to hepatic metastases

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* No chronic medical condition requiring treatment with corticosteroids
* No prior severe hypersensitivity reaction to agents containing Cremophor (polyoxyethylated castor oil)
* No serious uncontrolled medical disorder, active infection, or psychiatric disorder (e.g., dementia) that would preclude study
* No preexisting neurotoxicity grade 1 or greater
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No more than 2 prior chemotherapy regimens for metastatic disease
* No prior platinum or taxane therapy
* No other concurrent chemotherapy

Endocrine therapy:

* At least 2 weeks since prior hormonal therapy (except megestrol for anorexia/cachexia) and recovered
* At least 7 days since prior corticosteroids
* No concurrent corticosteroids
* No concurrent hormonal therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy to 30% or more of bone marrow and recovered
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No other concurrent investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Primary Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Sullivan, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Result] Fishman MN, Garrett CR, Simon GR, Chiappori AA, Lush RM, Dinwoodie WR, Mahany JJ, Dellaportas AM, Cantor A, Gollerki A, Cohen MB, Sullivan DM. Phase I study of the taxane BMS-188797 in combination with carboplatin administered every 3 weeks in patients with solid malignancies. Clin Cancer Res. 2006 Jan 15;12(2):523-8. doi: 10.1158/1078-0432.CCR-05-0928. PMID 16428495